CLINICAL TRIAL: NCT01940601
Title: An Open Label, Randomized, Active Controlled, Dose Finding Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Efficacy and Safety of Balugrastim at Doses of 300 µg/kg and 670 µg/kg in Pediatric Patients Diagnosed With Solid Tumors Receiving Chemotherapy
Brief Title: Pharmacodynamics, Pharmacokinetics, Efficacy and Safety of Balugrastim in Pediatric Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUGR-005
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Solid Tumors
Keywords: solid tumors; balugrastim
MeSH Terms: interventions — balugrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Balugrastim 300 ug/kg (Experimental): Balugrastim 300 μg/kg subcutaneously (SC) administration once per chemotherapy cycle, approximately 24 h after chemotherapy, up to 4 cycles
  Interventions: Drug: Balugrastim
- Balugrastim 670 μg/kg (Experimental): Balugrastim 670 μg/kg (maximum 40 mg) SC administration once per chemotherapy cycle, approximately 24 h after chemotherapy, up to 4 cycles
  Interventions: Drug: Balugrastim
- Filgrastim 5 μg/kg (Active Comparator): Filgrastim will be administered at a dose of 5 μg/kg SC once a day for at least 5 consecutive days or until absolute neutrophil count (ANC) has returned to ≥2*10^9/L for each chemotherapy cycle up to 4 cycles. The maximum period of filgrastim administration is 14 days in each cycle.
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Balugrastim — Balugrastim 300 ug/kg and Balugrastim 670 ug/kg
  Arms: Balugrastim 300 ug/kg; Balugrastim 670 μg/kg
Drug: Filgrastim — Filgrastim 5 μg/kg
  Arms: Filgrastim 5 μg/kg

SUMMARY:
The primary objective of this study is to find the optimal dose of balugrastim by characterizing its pharmacokinetics (PK), and by comparing the pharmacodynamics (PD) of balugrastim to filgrastim in children receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytologically-confirmed solid tumor in a patient for whom the study chemotherapy regimen [Vincristine plus ifosfamide plus doxorubicin plus etoposide (VIDE), Vincristine plus doxorubicin plus cyclophosphamide alternating with ifosfamide plus etoposide (VDC/IE), Ifosfamide plus vincristine plus actinomycin D (IVA) or Ifosfamide plus vincristine plus Adriamycin (IVAd)] is considered an appropriate treatment.
2. Minimum body weight of 15 kg
3. Life expectancy of at least 3 months with appropriate therapy
4. Female or male children and adolescents aged 2 to 17 years
5. Written informed consent provided by parent(s)/legal representative(s) of the pediatric patient and patient's assent if appropriate at the time of screening.
6. Fertile patients (male or female) must use highly reliable contraceptive measures.
7. Female patients who have attained menarche must have a negative urine pregnancy test at the screening visit.
8. White blood cell (WBC) count >2.5*10^9/L, ANC ≥1.5*10^9/L, and platelet count ≥100*10^9/L (at screening and prior to chemotherapy)

Exclusion Criteria:

1. Primary myeloid disorders
2. Prior radiation therapy within 4 weeks of randomization into this study.
3. Previous exposure to filgrastim, pegfilgrastim, lenograstim or other G-CSF less than 6 months before randomization.
4. Known hypersensitivity to filgrastim, pegfilgrastim, lenograstim or any balugrastim excipients
5. Pregnancy or breastfeeding (if a patient becomes pregnant during the study she will be withdrawn from the study).
6. Major surgery, serious infection, within 3 weeks before first administration of study drug, serious trauma or compound medical procedure within the 4 weeks prior to the first study drug dose.
7. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG, laboratory tests or imaging.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of absolute neutrophil count (ANC) | Day 1 to 14

SECONDARY OUTCOMES:
ANC nadir | Baseline to Week 16
  ANC nadir (measured in 10^9/L), which is the lowest ANC recorded
Time to ANC nadir | Baseline to Week 16
  Time to ANC nadir, which is the time from the beginning of chemotherapy up to the occurrence of the ANC nadir
Time to ANC recovery | Baseline to Week 16
  Time to ANC recovery (ANC >1.5*10^9/L) from nadir within each treatment cycle
Duration of severe neutropenia (DSN) | Baseline to Week 16
  Number of days subject experiences severe neutropenia (ANC <0.5*10^9/L)
Incidence of severe neutropenia | Baseline to Week 16
  Proportion of subjects who experience severe neutropenia (ANC <0.5*10^9/L)
Frequency of febrile neutropenia | Baseline to Week 16
  Frequency of febrile neutropenia (defined as body temperature >38.5°C for more than one hour [axillary measurement] and ANC <0.5*10^9/L) by cycle and across all cycles.
Summary of Participants with Adverse Events | From signing of informed consent to 16 weeks